CLINICAL TRIAL: NCT05721638
Title: Efficacy of Serum and Urinary Neutrophil Gelatinase-associated Lipocalin in the Early Detection of Acute Kidney Injury After Major Abdominal Surgery
Brief Title: Neutrophil Gelatinase-associated Lipocalin in Major Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Antalya Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Erhan Ozyurt, Associate Professor, Antalya Training and Research Hospital
Other Study IDs: Erhanter01
Record Dates: First submitted 2023-02-01; First posted 2023-02-10 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Acute Kidney Injury
Keywords: Acute Kidney Injury; Neutrophil gelatinase-associated lipocalin; Major abdominal surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Neutrophil gelatinase-associated lipocalin — Neutrophil gelatinase-associated lipocalin (NGAL) is a 25 KDa, neutrophil-derived molecule from the lipocalin family. It is also secreted in small amounts from kidney, prostate, and respiratory tract epithelial cells. After ischemic and nephrotoxic acute tubular necrosis, NGAL levels peak at the 3rd hour and remain elevated for approximately 24 hours. In patients who do not progress to AKI, NGAL levels begin to decrease as of the 1st hour after injury.

SUMMARY:
Acute kidney injury (AKI) after major surgery is a well-known complication. The incidence of AKI after major surgery ranges from 13% to 50%. The morbidity and mortality rates increase in patients with AKI due to the treatments applied and the prolonged hospital stay. In addition, as a result of all these processes, hospital costs increase and burden the health systems.

Classifications such as Acute Kidney Injury Network (AKIN) or Kidney Disease Improving Global Outcomes (KDIGO) are used in the diagnosis of AKI. In these classifications, evaluation is made based on kidney damage, serum creatinine (Scr), and urine output. However, Scr; is affected by factors such as age, gender, diet, muscle mass, and medication. In addition, in healthy individuals in terms of kidney reserve, a loss of up to 50% in nephrons is tolerated by the body and there is no change in Scr values. Therefore, the onset of the increase in Scr values occurs 48-72 hours after kidney damage. This situation causes delays in the treatments applied and increases morbidity and mortality rates.

For these reasons, interest in biomarkers used in the early diagnosis of AKI has increased in recent years. Neutrophil gelatinase-associated lipocalin (NGAL) is a 25 KDa, neutrophil-derived molecule from the lipocalin family. It is also secreted in small amounts from kidney, prostate, and respiratory tract epithelial cells. After ischemic and nephrotoxic acute tubular necrosis, NGAL levels peak at the 3rd hour and remain elevated for approximately 24 hours. In patients who do not progress to AKI, NGAL levels begin to decrease in the 1st hour after injury.

When the current literature is examined, scientific studies on NGAL have mostly been carried out on cardiovascular surgery cases to date. There are very few studies evaluating NGAL levels in patients who develop AKI after major abdominal surgery. These few studies evaluated either serum NGAL or urinary NGAL levels. In this study, both serum NGAL and urinary NGAL will be measured simultaneously to detect AKI that may develop in patients undergoing major abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III,
* Patients undergoing elective major abdominal surgery

Exclusion Criteria:

* Chronic renal failure,
* Using nephrotoxic drugs,
* Patients with a history of kidney transplantation or nephrectomy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who will undergo major abdominal surgery in Antalya Training and Research Hospital.
Sampling Method: Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Plasma NGAL Level | Postoperative 4th hour
  From patients undergoing major abdominal surgery, a blood sample will be taken at Postop 4th Hour for serum NGAL analysis.
Urine NGAL level | Postoperative 4th hour
  Urine samples will be collected from patients undergoing major abdominal surgery at the 4th postoperative hour for urine NGAL analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Erhan OZYURT, MD, Principal Investigator — Antalya Training and Research Hospital
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pan HC, Yang SY, Chiou TT, Shiao CC, Wu CH, Huang CT, Wang TJ, Chen JY, Liao HW, Chen SY, Huang TM, Yang YF, Lin HY, Chan MJ, Sun CY, Chen YT, Chen YC, Wu VC. Comparative accuracy of biomarkers for the prediction of hospital-acquired acute kidney injury: a systematic review and meta-analysis. Crit Care. 2022 Nov 12;26(1):349. doi: 10.1186/s13054-022-04223-6. PMID 36371256